CLINICAL TRIAL: NCT02564744
Title: A Phase 2 Study to Evaluate the Efficacy and Tolerability of Debio 1562 in Combination With Rituximab in Patients With Relapsed and/or Refractory Diffuse Large B-Cell Lymphoma and Other Forms of Non-Hodgkin's Lymphoma
Brief Title: Study to Evaluate the Efficacy and Tolerability of Debio 1562 in Combination With Rituximab in Participants With Relapsed and/or Refractory DLBCL and Other Forms of NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1562-201; 2015-004061-87 (EudraCT Number)
Record Dates: First submitted 2015-09-11; First posted 2015-10-01 (Estimated); Results first posted 2024-05-17 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Large B-Cell Lymphoma; B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: The interventional study model is sequential for Part 1 and Part 2/3 of the study, and parallel for Cohorts 1 and 2 of Part 1, and for Cohorts A and B of Part 2/3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Safety Run-in (Experimental): Participants with a diagnosis of relapsed and/or refractory (R/R) Diffuse Large B-Cell Lymphoma (DLBCL), and with non-Hodgkin's lymphoma (NHL) including follicular lymphoma (FL), marginal zone lymphoma/mucosa-associated lymphoid tissue (MZL/MALT), mantle cell lymphoma (MCL) or other NHL with the Sponsor's approval received Debio 1562 0.7 mg/kg, intravenous (IV) infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of 21-day cycles until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
  Interventions: Drug: Debio 1562; Drug: Rituximab
- Part 1: Cohort 1 (Experimental): Participants with R/R DLBCL received Debio 1562 0.7 mg/kg, IV infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of 21-day cycles until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
  Interventions: Drug: Debio 1562; Drug: Rituximab
- Part 1: Cohort 2 (Experimental): Participants with R/R, FL, MZL/MALT, MCL or other NHL with the Sponsor's approval received Debio 1562 0.7 mg/kg, IV infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of 21-day cycles until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
  Interventions: Drug: Debio 1562; Drug: Rituximab
- Part 2/3: Cohort A (Experimental): Participants with relapsed DLBCL received Debio 1562 0.7 mg/kg, IV infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of a 21-day cycle for at least 6 cycles and/or until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
  Interventions: Drug: Debio 1562; Drug: Rituximab
- Part 2/3: Cohort B (Experimental): Participants with relapsed DLBCL received Debio 1562 0.4 mg/kg IV infusion followed by rituximab 375 mg/m^2 IV infusion on Day 1, then Debio 1562 0.2 mg/kg IV infusion on Days 8 and 15 of a 21-day cycle for at least 6 cycles and/or until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
  Interventions: Drug: Debio 1562; Drug: Rituximab

INTERVENTIONS:
Drug: Debio 1562 — Administered as IV Infusion.
Drug: Rituximab — Administered as IV Infusion.

SUMMARY:
The primary purpose of the study was to determine the safety and tolerability, anti-tumor activity of the proposed Debio 1562 dose regimens in combination with rituximab.

ELIGIBILITY:
Inclusion Criteria:

* For Part 1 of the study, participants must have histopathologically confirmed diagnosis of R/R, DLBCL, FL, MZL/MALT, MCL, or other Sponsor approved NHL subtypes according to the World Health Organization (WHO) classification 2008 for which standard measures do not exist or are no longer effective.
* For Part 2 and Part 3 of the study, participants must have histopathologically and clinically confirmed diagnosis of relapsed DLBCL. Participants will be considered to have a relapsed disease if they showed a duration of response of at least 24 weeks after their first line of therapy. The following participants with relapsed DLBCL will be enrolled:

  1. Participants who received only one line of previous therapy and achieved either complete response (CR) or partial response (PR) for at least 24 weeks (from the last day of the last cycle) after their first line of therapy, but are not eligible for high dose chemotherapy with autologous stem cell transplantation (HD-ASCT)
  2. Participants who received more than one line of previous therapy (including HD-ASCT), and have achieved a duration of response (CR or PR) of at least 8 weeks (from the last day of the last cycle) after their last line of therapy
* Participants must have evaluable or measurable disease in accordance with the International Working Group Guidelines for Lymphoma.
* Participants must have received at least one but no more than six prior treatment regimens. Prior treatment with an anti-cluster of differentiation 20 (anti-CD20) agent, either alone or in combination, is allowed.
* Participants must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 2.
* Participants who are Hepatitis B surface antigen positive (HBsAg+) (must be polymerase chain reaction (PCR) negative) who are taking antivirals, are allowed to enroll.

Exclusion Criteria:

* Participants with a diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL).
* For Part 2 and Part 3 of the study, participants with primary refractory DLBCL (defined as progression of disease within 24 weeks after first line of treatment).
* For Part 2 and Part 3 of the study, participants that are eligible to undergo first time HD-ASCT.
* For Part 2 and Part 3 of the study, participants with R/R FL, MZL/MALT, MCL, or any other NHL subtypes according to the WHO classification.
* Participants with active hepatitis A, B or C infection.
* Women who are pregnant or breast feeding.
* Participants who have received prior therapy with other anti-CD37-targeting therapy.
* Participants who have known central nervous system, meningeal, or epidural disease including brain metastases.
* Participants with impaired cardiac function or clinically significant cardiac disease.
* Participants currently presenting interstitial lung disease, diffuse parenchymal lung disease, or with a past history of severe/Grade 3 parenchymal lung disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-05 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (9):
  - Alabama Oncology, Birmingham, Alabama
  - Carle Foundation Hospital, Cancer Center, Urbana, Illinois
  - Abbott Northwestern Hospital, Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Novant Health Oncology, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- Belgium (4):
  - CHU UCL Namur asbl - Site Godinne, Yvoir, Namur
  - Jan Yperman Ziekenhuis, Ieper, West-Vlaanderen
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
  - St. Augustinus Hospital, Department of Hematology, Wilrijk
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv
  - Specialized Hospital for Active Treatment of Hematological Diseases,Clinic of Hematology, Sofia
  - Multiprofile Hospital for Active Treatment - Hristo Botev, Vratsa, Vratsa
- Czechia (4):
  - University Hospital Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Kralovske Vinohrady, Prague
  - General University Hospital in Prague, Prague
- Hungary (3):
  - National Institute of Oncology, Budapest
  - University of Debrecen Clinical Center, Debrecen
  - Medical Center of the University of Pecs, Pécs
- Italy (4):
  - University Hospital - Ospedali Riuniti Umberto I - GM Lancisi - G Salesi of Ancona, Ancona
  - Civil Hospital of Brescia, Brescia
  - United Hospitals Villa Sofia Cervello, Palermo
  - Local Healthcare Company 8 Berica (Azienda ULSS8 Berica), Hospital San Bortolo of Vicenza, Vicenza
- Poland (4):
  - University Clinical Center in Gdansk, Gdansk
  - Provincial Hospitals in Gdynia Sp. z o.o. (LLC), Gdynia
  - Małopolskie Medical Centre, Krakow
  - St. John of Dukla Oncology Center of Lublin Land, Lublin
- Regional Hospital of Bellinzona and Valli, Oncology Institute of Southern Switzerland, Bellinzona, Canton Ticino, Switzerland
- Ukraine (7):
  - Cherkasy Regional Oncology Center, Regional Treatment and Diagnostic Hematology Center, Cherkasy
  - Grigoriev Institute for Medical Radiology and Oncology of the National Academy of Medical Sciences of Ukraine, Kharkiv
  - Communal Non-profit enterprise "Regional Center of Oncology", Kharkiv
  - National Institute of Cancer, Kyiv
  - National Research Center for Radiation Medicine, Kyiv
  - Kyiv City Clinical Hospital #9, City Hematology Center, Kyiv
  - Podillia Regional Oncology Center, Vinnytsia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 38 investigative sites in the United States, Belgium, Ukraine, the Czech Republic, Hungary, Bulgaria, Italy, Poland, and Switzerland from 05 June 2016 to 25 June 2021.
Pre-assignment Details: A total of 127 participants were screened and 100 participants with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) and other forms of non-Hodgkin's lymphoma (NHL) were enrolled, 37 participants into Part 1 and 63 participants into Part 2/3.
Groups:
- Part 1: Safety Run-in: Participants with a diagnosis of R/R DLBCL, and with NHL including follicular lymphoma (FL), marginal zone lymphoma/mucosa-associated lymphoid tissue (MZL/MALT), mantle cell lymphoma (MCL) or other NHL with the Sponsor's approval received Debio 1562 0.7 mg/kg, intravenous (IV) infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of 21-day cycles until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
Period: Overall Study
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Started | 17 | 8 | 12 | 33 | 30
Efficacy Evaluable (EE) Population (EE population included all participants who received at least one dose of Debio 1562 and rituximab and had both baseline and post-baseline evaluable disease assessments (including clinical progressive disease [PD]).) | 15 | 8 | 11 | 30 | 30
Pharmacokinetic (PK) Population (PK population included all participants who received at least one dose of Debio 1562 or rituximab and had at least one PK concentration result available.) | 17 | 8 | 12 | 32 | 29
Anti-drug Antibody (ADA) Population (ADA population included all participants who received at least one dose of Debio 1562 or rituximab and had at least one ADA post exposure result available.) | 14 | 6 | 10 | 30 | 25
Completed | 5 | 1 | 4 | 14 | 10
Not Completed | 12 | 7 | 8 | 19 | 20
Not completed — Investigator decision | 0 | 0 | 0 | 0 | 1
Not completed — Death | 10 | 5 | 4 | 16 | 16
Not completed — End of study Page Missing | 0 | 0 | 3 | 3 | 0
Not completed — Subject Withdrew Consent | 1 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 1
Not completed — Reason not specified | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants from the screened population who received at least one dose of Debio 1562.
Groups:
- Part 1: Safety Run-in: Participants with a diagnosis of R/R DLBCL, and with NHL including FL, MZL/MALT, MCL or other NHL with the Sponsor's approval received Debio 1562 0.7 mg/kg, IV infusion followed by rituximab 375 mg/m^2 IV infusion, once on Day 1 of 21-day cycles until the study discontinuation criteria were met (until they develop disease progression, death, unacceptable toxicity, withdraw consent, start new anti-lymphoma treatment or the Sponsor terminates the study).
- Total: Total of all reporting groups
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B | Total
Number analyzed (Participants) | 17 | 8 | 12 | 33 | 30 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (13.05) | 70.1 (9.79) | 68.5 (5.92) | 65.7 (13.26) | 68.7 (11.78) | 67.8 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 14 | 15 | 44
  Male | 12 | 3 | 7 | 19 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 2 | 5
  Not Hispanic or Latino | 15 | 5 | 12 | 32 | 28 | 92
  Unknown or Not Reported | 1 | 2 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1
  White | 16 | 7 | 11 | 31 | 30 | 95
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered study drug related. This included exacerbation of a pre-existing condition. AEs included worsening (change in nature, severity, or frequency) of conditions present at the onset of the study, intercurrent illnesses, drug interactions, events related to or possibly related to concomitant medications, abnormal laboratory values (this included significant shifts from baseline within the range of normal that the Investigator considered to be clinically important), clinically significant abnormalities in physical examination, vital signs, and weight.
Time Frame: Up to 30 days after end of treatment (EOT) (Up to 38 months)
Population: Safety population included all participants from the screened population who received at least one dose of Debio 1562.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 17 | 8 | 12 | 33 | 30
Participants | 16 | 8 | 12 | 32 | 29

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Test Results Reported as TEAEs
Description: The clinical laboratory tests included Hematology: Hematocrit (Hct), hemoglobin (Hgb), platelet count, red blood cell (RBC) count, white blood cell (WBC) count with differential; Serum Chemistry: Albumin (ALB), alkaline phosphatase (ALK-P), alanine aminotransferase (ALT), aspartate aminotransferase (AST), blood urea nitrogen (BUN), calcium (Ca), chloride (Cl), creatinine, glucose, lactate dehydrogenase (LDH), magnesium, phosphorus, potassium (K), sodium (Na), total bilirubin, total protein, uric acid, immunoglobulin levels (IgG, IgA, IgM); Urinalysis: Appearance, specific gravity and pH, evaluation of glucose, protein, bilirubin, ketones, leukocytes and blood; Coagulation: Prothrombin time (PT) or international normalized ratio (INR), activated partial thromboplastin time (aPTT).
Time Frame: Up to 30 days after EOT (Up to 38 months)
Population: Safety population includes all participants from the screened population who received at least one dose of Debio 1562.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 17 | 8 | 12 | 33 | 30
Participants
  Neutrophil Count Decreased | 6 | 1 | 2 | 2 | 2
  Lymphocyte Count Decreased | 5 | 1 | 0 | 0 | 0
  WBC Count Decreased | 5 | 0 | 0 | 1 | 3
  Platelet Count Decreased | 4 | 1 | 3 | 0 | 2
  Anaemia | 0 | 2 | 2 | 7 | 6
  Leukopenia | 0 | 1 | 1 | 5 | 7
  Neutropenia | 1 | 1 | 4 | 21 | 17
  Lymphopenia | 0 | 0 | 0 | 8 | 6
  Hypophosphataemia | 1 | 0 | 1 | 1 | 0
  Thrombocytopenia | 0 | 1 | 1 | 4 | 6
  Febrile Neutropenia | 2 | 0 | 1 | 1 | 1
  AST Increased | 2 | 2 | 1 | 0 | 1
  ALK-P Increased | 3 | 0 | 1 | 1 | 1
  ALT Increased | 2 | 1 | 0 | 1 | 1
  Blood Creatinine Increased | 0 | 1 | 1 | 1 | 0
  Hemoglobin Decreased | 2 | 0 | 0 | 0 | 0
  Blood Immunoglobulin G Decreased | 0 | 0 | 0 | 1 | 1
  Blood Magnesium Decreased | 0 | 0 | 0 | 0 | 0
  Hyperkalaemia | 1 | 1 | 2 | 0 | 2
  Hypoalbuminaemia | 0 | 0 | 0 | 2 | 0
  Hypercalcaemia | 1 | 0 | 0 | 2 | 1
  Hyperglycaemia | 0 | 0 | 0 | 2 | 0
  Hypernatraemia | 0 | 0 | 1 | 0 | 1
  Hyponatraemia | 2 | 0 | 0 | 0 | 1
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0
  Hyperuricaemia | 0 | 0 | 1 | 1 | 0
  Hypoglycaemia | 1 | 0 | 1 | 0 | 0
  Hypomagnesaemia | 0 | 0 | 1 | 1 | 0
  Blood Bilirubin Increased | 1 | 0 | 0 | 1 | 0
  Hypokalaemia | 2 | 0 | 2 | 0 | 2
  Gamma-glutamyl transferase Increased | 0 | 0 | 0 | 2 | 1

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Reported as TEAEs
Description: A standard 12-lead ECG was performed.
Time Frame: Up to 30 days after EOT (Up to 38 months)
Population: Safety population included all participants from the screened population who received at least one dose of Debio 1562.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 17 | 8 | 12 | 33 | 30
Participants
  Atrial Fibrillation | 0 | 0 | 1 | 0 | 1
  Electrocardiogram QT prolonged | 0 | 0 | 0 | 1 | 1
  Acute myocardial infarction | 1 | 0 | 1 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Sign Measurements Reported as TEAEs
Description: Vital signs included systolic and diastolic blood pressure, heart rate, temperature, and respiratory rate.
Time Frame: Up to 30 days after EOT (Up to 38 months)
Population: Safety population included all participants from the screened population who received at least one dose of Debio 1562.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 17 | 8 | 12 | 33 | 30
Participants
  Body Temperature Increased | 1 | 0 | 0 | 1 | 0
  Hypertension | 0 | 0 | 0 | 3 | 2
  Hypotension | 0 | 0 | 1 | 1 | 0
  Pyrexia | 4 | 2 | 1 | 6 | 4
  Hyperthermia | 0 | 0 | 0 | 0 | 2
  Tachycardia | 1 | 0 | 0 | 0 | 1

5. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a Best overall response (BOR) of partial response (PR) or complete response (CR). BOR was the best response recorded from the start of the treatment until disease progression, initiation of new anti-cancer therapy, or end of the study period, whichever occurred first. CR was defined as disappearance of all target lesions, no new lesions formation. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to ≤1.5 cm. PR was defined as ≥50% decrease in the sum of diameters of up to 6 target measurable nodes or extranodal sites, no new lesions formation.
Time Frame: Up to Progressive Disease (PD) or death (up to approximately 55 months) or initiation of new anti-cancer therapy whichever occurs first
Population: EE population included all participants who received at least one dose of Debio 1562 and rituximab and had both baseline and post-baseline evaluable disease assessments (including clinical PD).
Measure: Number (95% Confidence Interval); unit: percent responders
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 15 | 8 | 11 | 30 | 30
percent responders | 26.7 [7.8 to 55.1] | 12.5 [0.3 to 52.7] | 81.8 [48.2 to 97.7] | 50.0 [31.3 to 68.7] | 50.0 [31.3 to 68.7]

6. Secondary Outcome: Maximum Plasma Drug Concentration (Cmax) of Debio 1562 and Rituximab
Time Frame: Parts 1, 2/3: Pre and Post infusion: 5 min-Day (D) 1 of Cycles (C) 1-8 and 2 hours (h)-D1 of C1-2 (for Part 2/3), 24h-D2, 48h-D3 and D8, 15 of C1, 2; D1 of Month 37 (EOT) (rituximab only) and Month 38 (follow-up) (Cycle=21 days)
Population: PK population included all participants who received at least one dose of Debio 1562 or rituximab and had atleast one PK concentration result available. Number analyzed signifies the number of participants with available data at the specific timepoint.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 17 | 8 | 12 | 32 | 29
nanogram per milliliter (ng/ml)
  Debio 1562: Cycle 1 | 10005.9 (4147.35) | 9411.5 (7762.98) | 11821.2 (5456.11) | 15339.4 (3514.51) | 6612.4 (2315.16)
  Debio 1562: Cycle 2: number analyzed (Participants) | 14 | 6 | 7 | 29 | 24
  Debio 1562: Cycle 2 | 8697.9 (3540.53) | 7775.0 (2646.11) | 10521.4 (3448.39) | 13868.6 (4143.59) | 8465.5 (6553.50)
  Debio 1562: Cycle 3: number analyzed (Participants) | 10 | 4 | 9 | 18 | 19
  Debio 1562: Cycle 3 | 10600.0 (3879.40) | 11472.5 (3684.63) | 13682.2 (3093.84) | 14324.4 (5532.63) | 6824.0 (2911.62)
  Debio 1562: Cycle 4: number analyzed (Participants) | 9 | 3 | 9 | 16 | 17
  Debio 1562: Cycle 4 | 7787.8 (3334.11) | 9230.0 (1980.08) | 11703.3 (2284.15) | 12560.0 (4625.17) | 7122.9 (3084.39)
  Debio 1562: Cycle 5: number analyzed (Participants) | 7 | 2 | 8 | 14 | 16
  Debio 1562: Cycle 5 | 9744.3 (1816.91) | 9675.0 (1308.15) | 13220.0 (2049.06) | 13487.1 (4458.46) | 7305.0 (3089.01)
  Debio 1562: Cycle 6: number analyzed (Participants) | 6 | 2 | 8 | 14 | 14
  Debio 1562: Cycle 6 | 8050.0 (2418.64) | 10195.0 (3825.45) | 12983.8 (3182.10) | 13025.7 (5043.89) | 6904.3 (2516.11)
  Debio 1562: Cycle 7: number analyzed (Participants) | 5 | 1 | 7 | 0 | 0
  Debio 1562: Cycle 7 | 7908.0 (3111.60) | 9940.0 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. | 12600.0 (1803.70) |  |
  Debio 1562: Cycle 8: number analyzed (Participants) | 3 | 0 | 8 | 0 | 0
  Debio 1562: Cycle 8 | 2253.0 (2214.31) |  | 12501.3 (2658.79) |  |
  Debio 1562: Month 38: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Debio 1562: Month 38 |  |  |  |  | 15000.0 (NA) — Standard deviation (SD) cannot be calculated for 1 participant.
  Rituximab: Cycle 1: number analyzed (Participants) | 16 | 8 | 12 | 32 | 29
  Rituximab: Cycle 1 | 213287.4 (55735.54) | 207415.8 (67408.74) | 179430.7 (41213.48) | 170942.3 (28871.50) | 171006.4 (37226.83)
  Rituximab: Cycle 2: number analyzed (Participants) | 14 | 7 | 11 | 29 | 24
  Rituximab: Cycle 2 | 251697.6 (41113.07) | 214761.9 (40919.84) | 191988.5 (65788.33) | 205481.9 (43738.73) | 210563.7 (43723.39)
  Rituximab: Cycle 3: number analyzed (Participants) | 9 | 4 | 9 | 18 | 18
  Rituximab: Cycle 3 | 272302.8 (58497.66) | 213378.8 (36470.96) | 239380.8 (60127.34) | 218358.1 (49891.16) | 254760.9 (107449.36)
  Rituximab: Cycle 4: number analyzed (Participants) | 8 | 3 | 9 | 16 | 17
  Rituximab: Cycle 4 | 283067.9 (57414.89) | 198313.3 (79455.19) | 262263.9 (67895.19) | 236146.8 (63699.49) | 267141.2 (65390.99)
  Rituximab: Cycle 5: number analyzed (Participants) | 7 | 2 | 8 | 14 | 15
  Rituximab: Cycle 5 | 366032.9 (94593.53) | 156582.0 (82703.21) | 266406.1 (52480.70) | 282017.6 (66512.79) | 267163.1 (51180.64)
  Rituximab: Cycle 6: number analyzed (Participants) | 6 | 2 | 8 | 14 | 14
  Rituximab: Cycle 6 | 354142.7 (90095.73) | 200913.0 (130086.43) | 240735.0 (114120.93) | 294989.5 (82301.31) | 296240.1 (68962.34)
  Rituximab: Cycle 7: number analyzed (Participants) | 5 | 1 | 7 | 1 | 0
  Rituximab: Cycle 7 | 341761.4 (37261.58) | 179381.0 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. | 281045.9 (62528.32) | 114902.0 (NA) — Standard deviation (SD) cannot be calculated for 1 participant. |
  Rituximab: Cycle 8: number analyzed (Participants) | 3 | 0 | 8 | 0 | 0
  Rituximab: Cycle 8 | 379038.7 (83552.42) |  | 251326.4 (85797.08) |  |
  Rituximab: Month 37: number analyzed (Participants) | 9 | 4 | 8 | 13 | 14
  Rituximab: Month 37 | 77330.7 (34343.07) | 59503.5 (9683.76) | 53960.9 (61954.05) | 86046.4 (53904.82) | 73469.1 (47009.66)
  Rituximab: Month 38: number analyzed (Participants) | 12 | 5 | 7 | 20 | 20
  Rituximab: Month 38 | 107690.6 (56044.52) | 82585.0 (31312.62) | 78777.3 (72013.43) | 69646.9 (49779.31) | 79561.6 (55656.86)

7. Secondary Outcome: Area Under the Time-concentration Curve From Time 0 to t (AUC0-t) of Debio 1562 and Rituximab
Time Frame: Parts 1, 2/3: Pre-dose, post infusion-5 min on Day 1 of C 1-6, 5 min on Day 1 of C 7, 8 and 2 h on Day 1 of C 1, 2 (only for Part 2/3), 24 h on Day 2, 48 h on Day 3, Days 8 and 15 of C 1, 2 (Cycle=21 days); EOT (up to 37 months), 30-day follow up
Population: Debio 1562 PK analysis was performed by population PK approach, this data was not collected. This data was also not collected for Rituximab.
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Area Under the Time-concentration Curve From Time 0 to Infinity (AUC0-inf) of Debio 1562 and Rituximab
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Terminal Half-life (t1/2) of Debio 1562 and Rituximab
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Clearance (CL) of Debio 1562 and Rituximab
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Debio 1562 and Rituximab
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Debio 1562 and Rituximab
Time Frame: as for outcome 7
Population: as for outcome 7
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the duration between the first dose date of Debio 1562 and the date of progressive disease (PD) or death due to any cause, whichever occurs first. PD is defined as the new or clear progression of preexisting non-measured lesions or regrowth of previously resolved lesions or a new node >1.5 cm in any axis or an abnormal lesion with >1.5 cm longest transverse diameter or increase by >50% of lesion.
Time Frame: Up to PD or death or end of study (approximately 57 months) or initiation of new anti-cancer therapy whichever occurs first
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 15 | 8 | 11 | 30 | 30
months | 1.4 [1.2 to 11.1] | 1.8 [1.3 to 4.0] | 20.7 [10.5 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to the low number of participants with events. | 5.1 [1.4 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to the low number of participants with events. | 4.6 [1.4 to 13.4]

14. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the duration between the first dose date of Debio 1562 and the date of first objective response (PR or CR). CR was defined as disappearance of all target lesions, no new lesions formation. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to ≤ 1.5 cm. PR was defined as ≥50% decrease in the sum of diameters of up to 6 target measurable nodes or extranodal sites, no new lesions formation.
Time Frame: as for outcome 13
Population: EE population included all participants who received at least one dose of Debio 1562 and rituximab and had both baseline and post-baseline evaluable disease assessments (including clinical PD). Overall number of participants analyzed signifies the number of participants who responded.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 4 | 1 | 9 | 15 | 15
months | 1.4 [1.2 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events. | 1.4 [NA to NA] — Lower and upper limits of 95% CI was not estimable due to the low number of participants with events. | 1.4 [1.4 to 2.1] | 1.5 [1.4 to 1.8] | 1.5 [1.4 to 3.3]

15. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as duration between date of the first objective response (PR or CR) and date of PD or death due to any cause, whichever occurs first. CR: Disappearance of all target lesions, no new lesions formation, any pathological lymph nodes (whether target or non-target) must have reduction in short axis to ≤1.5 cm. PR: ≥50% decrease in sum of diameters of up to 6 target measurable nodes or extranodal sites, no new lesions formation. PD: New or clear progression of preexisting non-measured lesions or regrowth of previously resolved lesions or a new node >1.5 cm in any axis or an abnormal lesion with >1.5 cm longest transverse diameter or increase by >50% of lesion.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 4 | 1 | 9 | 15 | 15
months | NA [9.7 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants with events. | 2.6 [NA to NA] — Lower and upper limits of 95% CI was not estimable due to the low number of participants with events. | NA [13.2 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants with events. | NA [13.6 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants with events. | 16.5 [3.4 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events.

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration between the first dose date of Debio 1562 and the date of death due to any cause.
Time Frame: Up to death or end of study (approximately 57 months) or one year from the last participant's first dose
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 15 | 8 | 11 | 30 | 30
months | 30.0 [13.3 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events. | 8.4 [2.7 to 17.0] | 34.3 [24.3 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events. | NA [11.4 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants with events. | 17.3 [9.5 to NA] — Upper limit of 95% CI was not estimable due to the low number of participants with events.

17. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) for Debio 1562
Description: The potential immunogenicity against Debio 1562 was assessed in an ADA population.
Time Frame: Part 1: Pre-dose on Day 1 of Cycle(C)1 to 8; Part 2/3: Pre-dose on Day 1 of C1 to 6 and on Day 1 of C7 for participants who received treatment beyond C6 (each C=21 days); Parts 1, 2/3: Month 37 (EOT) and Month 38 (30-Day FU visit) (Cycle=21 days)
Population: ADA population included all participants who received at least one dose of Debio 1562 or rituximab and had at least one ADA post exposure result available. Overall number of participants analyzed signifies number of participants with non-missing ADA value at baseline and at least one non-missing post-treatment value.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
Number analyzed (Participants) | 14 | 6 | 10 | 30 | 25
Participants
  No Change From Baseline | 13 | 6 | 10 | 25 | 20
  Decrease in ADA Titer From Baseline | 1 | 0 | 0 | 3 | 3
  Increase in ADA Titer From Baseline | 0 | 0 | 0 | 2 | 2

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to end of study (approximately 57 months); Adverse events: Up to 30 days after EOT (Up to 38 months)
Description: Safety Population included all participants from the screened population who received at least 1 dose of Debio 1562.
Arm/Group | Part 1: Safety Run-in | Part 1: Cohort 1 | Part 1: Cohort 2 | Part 2/3: Cohort A | Part 2/3: Cohort B
All-Cause Mortality (participants affected / at risk) | 11/17 | 6/8 | 5/12 | 16/33 | 17/30
Serious Adverse Events (participants affected / at risk) | 5/17 | 3/8 | 5/12 | 15/33 | 9/30
Other Adverse Events (participants affected / at risk) | 15/17 | 8/8 | 12/12 | 32/33 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Safety Run-in (N=17) | Part 1: Cohort 1 (N=8) | Part 1: Cohort 2 (N=12) | Part 2/3: Cohort A (N=33) | Part 2/3: Cohort B (N=30)
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Circulatory collpase (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis aspergillus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Safety Run-in (N=17) | Part 1: Cohort 1 (N=8) | Part 1: Cohort 2 (N=12) | Part 2/3: Cohort A (N=33) | Part 2/3: Cohort B (N=30)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 3 | 2
Flushing (Vascular disorders) | 0 | 0 | 2 | 1 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Lymphostasis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Cyanosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Malignant muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 1 | 4 | 7 | 2
Pyrexia (General disorders) | 4 | 2 | 1 | 6 | 4
Asthenia (General disorders) | 1 | 1 | 4 | 0 | 5
Oedema peripheral (General disorders) | 0 | 0 | 4 | 0 | 2
Chills (General disorders) | 1 | 0 | 2 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 2 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 6 | 1 | 2 | 2 | 2
Lymphocyte count decreased (Investigations) | 5 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 5 | 0 | 0 | 1 | 3
Platelet count decreased (Investigations) | 4 | 1 | 3 | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 1 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 21 | 17
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 5 | 7
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 7 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 4 | 6
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 6 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 5 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 4 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5 | 5 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 4 | 2 | 4
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 6
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Lividity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Iliolumbar syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1 | 1 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 3 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 2 | 4 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis aspergillus (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once an agreement between the Sponsor and the Investigator has been reached.

DOCUMENTS (2):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT02564744/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT02564744/SAP_001.pdf